CLINICAL TRIAL: NCT01817946
Title: Myotubular Myopathy Genetic Testing Study
Status: Completed | Type: Observational
Sponsor: Cure CMD (Other)
Collaborators: Valerion Therapeutics, LLC (Industry); Congenital Muscle Disease International Registr (Other); University of Chicago (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMDIR-001
Record Dates: First submitted 2013-03-19; First posted 2013-03-26 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Myotubular Myopathy
Keywords: Congenital Myopathy; Centronuclear Myopathy; Myotubular Myopathy; Myotubularin; MTM1 Gene; Genetic testing; Sequencing; Deletion/Duplication Mutation; CGH array
MeSH Terms: conditions — Myopathies, Structural, Congenital; Myotonia Congenita | interventions — Genetic Testing; Base Sequence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva, whole blood, or other source
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Genetic testing: All participants determined eligible for the study will be placed into genetic testing arm.
  Interventions: Other: Genetic Testing

INTERVENTIONS:
Other: Genetic Testing — Genetic testing services will be provided by the University of Chicago under the guidance of Dr. Soma Das, PhD. Services will be coordinated by Rachel Alvarez, CMDIR Associate Director. Genetic testing will include standard sequencing of the MTM1 gene followed by CGH array for deletion/duplication in cases where no pathologic variant is identified by standard sequencing.
  Other Names: Sequencing

SUMMARY:
Myotubular myopathy (XLMTM) is an X-linked disorder caused by mutations in the myotubularin gene (MTM1). The clinical spectrum is variable and ranges from individuals who require a wheelchair and full time breathing support to those who are able to walk and breathe on their own. Symptoms of myotubular myopathy include long faces, facial weakness with eye muscle weakness, breathing support with a muscle biopsy demonstrating central nucleated fibers. These symptoms may be caused by mutations or changes in the MTM1, BIN1 (bridging integrator 1), DNM2 (dynamin 2) and RYR1 (ryanodine receptor 1) genes. However, the majority are caused by mutations in the MTM1 gene. Some patients with symptoms consistent with myotubular myopathy who initially have negative testing of the MTM1 gene were later found to have a unique type of change in the MTM1 gene. This unique change, called a deletion or duplication, can be found with a different type of genetic test called a CGH (comparative genomic hybridization) array.

Investigators do not know how frequent deletions and duplications are in patients with X-linked myotubular myopathy. Recently, there have been advances in identifying potential treatments for XLMTM. The next step will be to proceed with clinical trials of potential treatments. In order to be ready for clinical trials, it is important that investigators find the specific genetic change that is causing XLMTM in people with this diagnosis. This study will attempt to find changes in the MTM1 gene in individuals who have clinical symptoms consistent with a diagnosis of XLMTM. Participants will be asked to enroll in the CMDIR (Congenital Muscle Disease International Registry), complete a brief clinical survey, provide access to medical records, and provide a saliva or blood sample for genetic testing. Results of genetic testing will be communicated to participants by the physician specified in the consent by the signing person.

Study Hypothesis:

Not all individuals with a clinical diagnosis of XLMTM have access to genetic testing. Investigators know that deletions and duplications of the MTM1 gene can cause XLMTM. Investigators will find more individuals with XLMTM by performing genetic testing of the MTM1 gene, including CGH array for deletions and duplications.

DETAILED DESCRIPTION:
* Prospective participants will complete registration in the CMDIR.
* The CMDIR genetic curator will review CMDIR data for study eligibility.
* If eligible, participant will be called and consented to participate in the study.
* Sequencing can be done with a saliva sample. However, if this method does not detect a mutation or change in the MTM1 gene, a further test, called CGH Array, has to be performed. For the CGH Array test, a saliva sample may deliver a clear result in terms of a deletion/duplication mutation. In the event, CGH Array with the saliva sample does not provide a result, a the blood sample is necessary to repeat CGH Array.
* The study participant will receive a kit and instructions for saliva specimen collection for genetic testing from the CMDIR in the mail.
* If a mutation or change in the MTM1 gene could not be found by genetic testing and CGH Array with a saliva sample, the study participant will receive a second kit in the mail from the CMDIR with instructions for a blood draw to be used for CGH Array.
* The family will coordinate collection of the saliva specimen or a local blood draw, if necessary, and will be responsible for mailing the specimen in a pre-paid parcel to the University of Chicago. There will be a $40 reimbursement for the cost of the blood draw. Mailing the specimen to the testing site is at no cost for the participant. A two-week turn-around from receipt of the kit to sending it to the testing laboratory is requested.
* Genetic testing will start with standard sequencing of the MTM1 gene, isolated from the saliva specimen, followed by CGH Array if sequencing of the MTM1 gene isolated from the saliva sample or further from a blood sample if a variant consistent with the symptoms could not be detected using the saliva sample.
* Test results will be 1) reported to a physician specified by the study participant and 2) uploaded into the study participant's profile in the CMDIR and 3) if concurrently enrolled in the Beggs Laboratory or other IRB-approved clinical study, test results will also be made available to that study provided appropriate informed consent has been given.

ELIGIBILITY:
Inclusion Criteria: Patient eligibility will be determined by the CMDIR genetic curator using the following prioritization protocol.

1. Males and females in the US and Canada who have a known mutation in the MTM1 gene identified in a research lab and never confirmed in a clinical CLIA (Clinical Laboratory Improvement Amendments) -certified laboratory.
2. Male and female patients in the US and Canada who meet 2 of 3 of the following criteria: + clinical history, + family history, + centronucleation on muscle biopsy (no signs of nemaline rods or cores). Clinical history includes: post-natal breathing support (not necessarily continued after first month), length above 90% for EGA (estimated gestational age), facial characteristics (narrow facies), facial weakness (ophthalmoplegia, excessive saliva with need for suctioning).
3. Males and females in the US and Canada who present with XLMTM symptoms and no genetic mutation in the MTM1 gene found with conventional sequencing, requiring CGH array deletion/duplication testing.
4. Age range: One month - no maximum age.
5. Individual is registered with the CMDIR.
6. Written study consent provided by parent/caregiver (affected individual's age less than 18 years or for those individuals greater than 18 years with learning disabilities or inability to physically access consent) or affected individual (age greater than 18 years)

Exclusion Criteria:

1. Carrier testing for asymptomatic mothers.

Min Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be composed of individuals registered in the CMDIR who have been clinically diagnosed with XLMTM but do not have an XLMTM diagnosis confirmed by genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Description of Mutations in the MTM1 Gene by Complete Genetic Sequencing | 1 year
  To confirm presence, locations and frequencies of mutations in the MTM1 gene in study participants presenting with symptoms as listed in the Brief Summary and muscle biopsy and/or family history typical for myotubular myopathy or prior confirmation of a mutation in the MTM1 gene by research sequencing.

SECONDARY OUTCOMES:
Frequency of Deletion/Duplication Mutations in the MTM1 Gene by CGH Array Testing | 1 year
  To establish the frequency of deletions/duplications in the MTM1 gene for patients who have negative sequencing but have clinical history/muscle biopsy/family history.
To Examine the Relation of the Mutation in the MTM1 Gene to the Phenotype | 2 years
  Investigators will compare mutations characterized by sequencing and CGH array (if necessary) with the following data in the study participant's CMDIR profile: age of onset, ventilatory support needed post-natal and ongoing, maximal motor function achieved, current motor function, need for gastrostomy tube and rate of ER visits and hospitalizations. The individual genotype - phenotype relation will then be compared to that of other study participants. In the event that a genotype-phenotype pattern can be established, this may help predict the course of the disease and prepare for appropriate care.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine de Chastonay, PhD, Principal Investigator — CMDIR; Elizabeth DeChene, MS, GCG, Principal Investigator — Children's Hospital of Philadelphia; Soma Das, PhD, Principal Investigator — University of Chicago Genetic Testing Services Laboratory
Locations (1):
- Congenital Muscle Disease International Registry, Torrance, California, United States

REFERENCES:
- [Background] Trump N, Cullup T, Verheij JB, Manzur A, Muntoni F, Abbs S, Jungbluth H. X-linked myotubular myopathy due to a complex rearrangement involving a duplication of MTM1 exon 10. Neuromuscul Disord. 2012 May;22(5):384-8. doi: 10.1016/j.nmd.2011.11.004. Epub 2011 Dec 9. PMID 22153990
- [Background] Oliveira J, Oliveira ME, Kress W, Taipa R, Pires MM, Hilbert P, Baxter P, Santos M, Buermans H, den Dunnen JT, Santos R. Expanding the MTM1 mutational spectrum: novel variants including the first multi-exonic duplication and development of a locus-specific database. Eur J Hum Genet. 2013 May;21(5):540-9. doi: 10.1038/ejhg.2012.201. Epub 2012 Sep 12. PMID 22968136
- [Background] Bevilacqua JA, Bitoun M, Biancalana V, Oldfors A, Stoltenburg G, Claeys KG, Lacene E, Brochier G, Manere L, Laforet P, Eymard B, Guicheney P, Fardeau M, Romero NB. "Necklace" fibers, a new histological marker of late-onset MTM1-related centronuclear myopathy. Acta Neuropathol. 2009 Mar;117(3):283-91. doi: 10.1007/s00401-008-0472-1. Epub 2008 Dec 16. PMID 19084976
- [Background] Gurgel-Giannetti J, Zanoteli E, de Castro Concentino EL, Abath Neto O, Pesquero JB, Reed UC, Vainzof M. Necklace fibers as histopathological marker in a patient with severe form of X-linked myotubular myopathy. Neuromuscul Disord. 2012 Jun;22(6):541-5. doi: 10.1016/j.nmd.2011.12.005. Epub 2012 Jan 20. PMID 22264517
- [Background] North KN. Clinical approach to the diagnosis of congenital myopathies. Semin Pediatr Neurol. 2011 Dec;18(4):216-20. doi: 10.1016/j.spen.2011.10.002. PMID 22172416
- [Background] Dowling JJ, Lawlor MW, Das S. X-Linked Myotubular Myopathy. 2002 Feb 25 [updated 2018 Aug 23]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1432/ PMID 20301605
- [Result] Tosch V, Vasli N, Kretz C, Nicot AS, Gasnier C, Dondaine N, Oriot D, Barth M, Puissant H, Romero NB, Bonnemann CG, Heller B, Duval G, Biancalana V, Laporte J. Novel molecular diagnostic approaches for X-linked centronuclear (myotubular) myopathy reveal intronic mutations. Neuromuscul Disord. 2010 Jun;20(6):375-81. doi: 10.1016/j.nmd.2010.03.015. PMID 20434914
- See also: Congenital Muscle Disease International Registry — https://www.cmdir.org